CLINICAL TRIAL: NCT04306679
Title: Assessing the Effects of Educational Training Aimed to Improve Pain-reporting Reliability in Children After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0091-19-RMB
Record Dates: First submitted 2020-03-08; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): The intervention, which was aimed to educate children on how to use pain scales and provide reliable pain assessments was based on a two short animation clips, lasting approximately 5 min each, and a short (5 min) guided interaction between the study nurse and the participants, in between the two clips.
  Interventions: Other: Animation clips
- Control (Other): Children underwent the routine pre-operative preparations, which included a section on pain assessment.
  Interventions: Other: Instructions

INTERVENTIONS:
Other: Animation clips — The first animation clip focuses on the importance of pain assessment introduce three pain scales (categorical, NPS and faces) followed by explanations on their properties and on the appropriate way to use them.The second movie was aimed to provide an opportunity to implement the new knowledge in case studies
  Arms: Interventional arm
Other: Instructions — Routine preoperative preparations, which included a section on pain assessment instructions.
  Arms: Control

SUMMARY:
Treating pain, just as treating other medical conditions, depends on accurate assessment of patient's condition. When assessing pain, as other subjective symptoms, the challenge is twofold because the assessment is dependent on patient's understanding and use of the scale, all the more so in children

So far, attempts to improve pain assessments have been focused on the development and refining pain scales. No emphasis has been placed on improving patient's ability to report their pain. Our purpose is to evaluate a training program designed to improve the quality of children's post-surgical pain intensity reports.

After receiving Helsinki approval, eligible children and their parents will signed informed-consent. After surgery, the children, their parents, and the department nurses will assess children's pain intensity. Immediately after the nurse assessment, parents will assess their child's pain (blindly and independently) and the children will report their pain on four different pain scales.

Children aged 8-17, hospitalized in Rambam medical-center for elective surgery will be invited to participate. Children in the experimental group will be exposed to a training program, developed for this study, aimed to teach and train how to report pain. The control group will receive the standard pre-surgical instructions.

ELIGIBILITY:
Inclusion Criteria:

1. children at age 8-17 years;
2. absence of psychiatry, cognitive, and/or neurological disorders;
3. understand the purpose and the instructions of the study, agree to participate and parent signed inform consent.

Exclusion Criteria:

1. children suffering from Post traumatic stress disorder.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Quality of pain intensity scores based on the concordance between pain reports on different scales. | Pain intensity rating before analgesic consumption.
  The average difference between scores reported on the different scales was calculated as follows: The difference between to pain scores reported on each possible pairs of two scales was calculated in absolute values. The average difference of the 6 pairs was calculated. The 5-point CAT was transformed into a 0-10 scale by multiplying its values by 2.5.
Quality of pain intensity scores based on the concordance between pain reports on different scales. | Pain intensity rating one hour after analgesic consumption.
  The average difference between scores reported on the different scales was calculated as follows: The difference between to pain scores reported on each possible pairs of two scales was calculated in absolute values. The average difference of the 6 pairs was calculated. The 5-point CAT was transformed into a 0-10 scale by multiplying its values by 2.5.

SECONDARY OUTCOMES:
The difference between children assessment vs. nurses assessment. | NPS ratings before and one hour after analgesic consumption
  The difference between children pain assessment vs. nurses assessment on a 0-10 numerical pain scale (NPS), in which 0 indicates "no pain" and 10 "the worst pain imaginable."
The average difference between children assessment vs. parents. | NPS ratings before and one hour after analgesic consumption
  The difference between children pain assessment vs. parents assessment on a 0-10 numerical pain scale (NPS), in which 0 indicates "no pain" and 10 "the worst pain imaginable."
The average decrease in pain following analgesia: NPS | NPS ratings before and one hour after analgesic consumption
  The average decrease in pain following analgesic consumption (Delta NPS) based on a 0-10 numerical pain scale (NPS), in which 0 indicates "no pain" and 10 "the worst pain imaginable."
Quality of pain intensity scores based on the concordance between pain reports on different scales. | Pain intensity ratings before analgesic consumption.
  The within-subjects standard deviation (SD) between the 4 pain scores (provided at the same time of assessment). To assure that variability will be appropriately reflected by this measure, subjects who reported only "0" or only "10" in all 4 scales were excluded from this analysis due to potential bias of the within-subjects SD due to floor or ceiling effects.
Quality of pain intensity scores based on the concordance between pain reports on different scales. | Pain intensity ratings one hour after analgesic consumption.
  The within-subjects standard deviation (SD) between the 4 pain scores (provided at the same time of assessment). To assure that variability will be appropriately reflected by this measure, subjects who reported only "0" or only "10" in all 4 scales were excluded from this analysis due to potential bias of the within-subjects SD due to floor or ceiling effects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, The Clinical Pain Innovation Lab, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zontag D, Kuperman P, Honigman L, Treister R. Agreement between children's, nurses' and parents' pain intensity reports is stronger before than after analgesic consumption: Results from a post-operative study. Int J Nurs Stud. 2022 Jun;130:104176. doi: 10.1016/j.ijnurstu.2022.104176. Epub 2022 Jan 15. PMID 35395574